CLINICAL TRIAL: NCT06776081
Title: Adipocyte-Derived Extracellular Vesicles; Novel Biomarker and Mediator of Obesity-Related Endothelial Dysfunction
Brief Title: Adipocyte-Derived Extracellular Vesicles, Weight Loss, and Endothelial Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Christopher DeSouza, Professor of Distinction, University of Colorado, Boulder
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 24-0523; 24TPA1301309 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Weight Loss
Keywords: Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Intervention: Phase 1 (No Intervention): Phase 1 is a cross-sectional study to compare whether circulating Ad-EVs are associated with obesity-related endothelial dysfunction in normal weight adults and adults with obesity.
- Experimental: Phase 2 (Experimental): Phase 2 employs an intervention study design, to determine in adults with obesity, the effects of intentional weight loss (12-weeks) on circulating Ad-EVs and their effect on endothelium-dependent vasodilation.
  Interventions: Other: Weight loss without pharmacotherapy

INTERVENTIONS:
Other: Weight loss without pharmacotherapy — Adults with obesity participating in the 12-week hypocaloric diet-induced weight loss intervention will be individually counseled by the Clinical and Translational Research Center (CTRC) bionutritionist to consume a hypocaloric diet consistent with current dietary recommendations for weight loss until a 6-10% weight loss is achieved.
  Arms: Experimental: Phase 2

SUMMARY:
Changes in adipose tissue biology are now recognized as a key factor underlying the increased risk of metabolic and cardiovascular disease with obesity. Clinical interest in adipocyte-derived extracellular vesicles (Ad-EVs) has intensified due to their potential as circulating biomarkers of adipose tissue health and systemic messengers, regulators and mediators of cardiometabolic health and disease with obesity.

The investigators hypothesize that elevated Ad-EVs in adults with obesity will be negatively associated with endothelium-dependent vasodilation. Furthermore, the investigators hypothesize that in adults with obesity, intentional weight loss-induced reduction in circulating Ad-EVs is associated with greater endothelium-dependent vasodilation.

ELIGIBILITY:
Inclusion criteria:

* Age ≥40 years
* BMI <25 kg/m2 and BMI >25 kg/m2 for Phase 1 and BMI >25 kg/m2 for Phase 2. Rationale for defining obesity as BMI >25 kg/m2

Exclusion criteria:

* Current smoker
* Chronic overt medical condition (e.g., evidence of coronary artery disease on resting ECG, any history of myocardial infarction or stroke, or cancer, diabetes based on fasting blood glucose concentration)
* Alcohol abuse or dependence defined as more than 14 standard drinks/week and no more than 4 standard drinks/day for men and 7 standard drinks/week and 3 standard drinks/day for women (a standard drink is defined as 12 ounces of beer, 5 ounces of wines, 1 ½ ounces of 80-proof distilled spirits) reported during the medical history/physical exam
* Stage III hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg)
* Regular vigorous aerobic/endurance exercise (>3 bouts/week, >30 minutes/bout at a workload >6 METS)
* Women who are pregnant or breastfeeding
* History of anaphylaxis to betadine, lidocaine, iodine
* Raynaud's disease
* History of clotting disorders
* Anyone taking blood thinners and clotting medications
* Anyone taking statin medication
* Planned pregnancy in coming 4-6 months

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Circulating adipocyte-derived extracellular vesicles (Ad-EVs) | Circulating Ad-EVs will measured during Phase 1 visit 2 which is ~2 weeks from their respective start date.
  Circulating Ad-EVs will be determined from a peripheral blood sample in normal weight and obese adults. Ad-EVs will be determined using flow cytometry. The samples will be incubated with perilipin A. Ad-EVs will be defined as perilipin A positive cells ranging in size 0.2-0.8 um.
Phase 2: Circulating adipocyte-derived extracellular vesicles (Ad-EVs) | Circulating Ad-EVs will be measured during Phase 2 visit 15 which is ~17 weeks from their respective start date.
  Circulating Ad-EVs will be determined from a peripheral blood sample following the obese participants 12-week weight loss intervention.
Phase 1: Forearm Blood Flow (FBF) Response to Acetylcholine (ACh) | FBF response to ACh will be measured during Phase 1 and the participant's visit 2 which is ~ 2 weeks from their respective start date.
  FBF is measured via strain-gauge venous occlusion plethysmography in response to saline for 5 minutes and then to ACh (4.0, 8.0 and 16.0 ug/100 mL tissue/min; the doses of ACh infused into the brachial artery) for 5 minutes at each dose. Flows during the last minute of saline and each drug dose are measured and the mean value reported.
Phase 2: Forearm Blood Flow (FBF) Response to Acetylcholine (ACh) | FBF response to ACh will be measured during Phase 2 and the participant's visit 15 which is ~17 weeks from their respective start date.
  FBF is measured via strain-gauge venous occlusion plethysmography in response to saline for 5 minutes and then to ACh (4.0, 8.0 and 16.0 ug/100 mL tissue/min; the doses of ACh infused into the brachial artery) for 5 minutes at each dose. Flows during the last minute of saline and each drug dose are measured and the mean value reported.
Phase 1: Forearm Blood Flow (FBF) Response to Sodium Nitroprusside (NTP) | FBF response to NTP will be measured during Phase 1 and the participant's visit 2 which is ~ 2 weeks from their respective start date.
  FBF is measured via strain-gauge venous occlusion plethysmography in response to saline for 5 minutes and then to NTP (1.0, 2.0 and 4.0 ug/100 mL tissue/min; the doses of NTP infused into the brachial artery) for 5 minutes at each dose. Flows during the last minute of saline and each drug dose are measured and the mean value reported.
Phase 2: Forearm Blood Flow (FBF) Response to Sodium Nitroprusside (NTP) | FBF response to NTP will be measured during Phase 2 and the participant's visit 15 which is ~17 weeks from their respective start date.
  FBF is measured via strain-gauge venous occlusion plethysmography in response to saline for 5 minutes and then to NTP (1.0, 2.0 and 4.0 ug/100 mL tissue/min; the doses of NTP infused into the brachial artery) for 5 minutes at each dose. Flows during the last minute of saline and each drug dose are measured and the mean value reported.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher DeSouza, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- University of Colorado Boulder Clinical and Translational Research Center (CTRC), Boulder, Colorado, United States